CLINICAL TRIAL: NCT04669639
Title: A Comparison of Erector Spinae Plane Block to Suprascapular Nerve Block for Analgesia in Shoulder Surgery
Brief Title: A Comparison of ESP Block to SSN Block for Analgesia in Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Naglaa Fathy Abdelhaleem Abdelhaleem, Lecturer, Anesthesia and Surgical Intensive Care department, Faculty of Medicine, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: #6506
Record Dates: First submitted 2020-11-25; First posted 2020-12-17 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2020-11

CONDITIONS: Arthroscopic Shoulder Surgery
Keywords: erector spinae plane block- suprascapular nerve

STUDY DESIGN:
Intervention Model Description: There has been a recent renewed interest in using the suprascapular nerve block (SSNB) as a phrenic nerve sparing approach for analgesia after shoulder surgery. The suprascapular nerve provides 70% of the sensory input to the glenohumeral joint and also innervates the infraspinatus and supraspinatus muscles. However, some researchers suggest that SSNB alone cannot provide a sufficient analgesia.The high-thoracic erector spinae plane block (HT-ESPB) has been described in several case reports as an effective analgesic modality for the shoulder region without causing motor or phrenic nerve block
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The care provider and outcome assessor will be unaware of the study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The block group (a) (Experimental): Patients were randomized in a 1:1 :1ratio, group (a) will receive SSN. The nerve blocks The procedure will be performed after induction of anaesthesia and endotracheal intubation.
  Interventions: Other: Block procedures for shoulder surgery analgesia
- The block group (b) (Experimental): Patients were randomized in a 1:1:1 ratio. group (b) will receive the Erector spinae plane block. The procedure will be performed after induction of anesthesia and endotracheal intubation.
  Interventions: Other: Block procedures for shoulder surgery analgesia
- control group (Placebo Comparator): Patients were randomized in a 1:1:1 ratio. this group will receive general anesthesia (GA) only
  Interventions: Other: Block procedures for shoulder surgery analgesia

INTERVENTIONS:
Other: Block procedures for shoulder surgery analgesia — The patients in group (a) will be placed in lateral decubitus. Then, an ultrasound-guided aseptic technique with a high-frequency linear transducer will be used to locate the transverse process of T2, where a needle will be inserted in a cephalocaudal direction until reaching the space between the fascia of the erector spinae and the transverse process of T2 and 30 ml of local anesthetic of bupivacaine 0.5% will be injected.
  * In group (b), SSC nerve block will be done as follow: In the suprascapular notch, an ultrasound-guided aseptic technique with a high-frequency linear transducer will be used. The linear probe, enveloped in a sterile sheath, will be placed parallel to the spine of the scapula to visualize it and then will be moved cephalic to the supraspinatus fossa. The probe will then be moved laterally up to the scapular notch, where the nerve will be identified by its round hyperechogenic shape 4 cm deep.
  * control group: patients will receive only general anesthesia

SUMMARY:
A comparison between Erector Spinae Plane block and Suprascapular nerve block in providing analgesia for shoulder surgery

DETAILED DESCRIPTION:
Suprascapular nerve block is considered a phrenic nerve sparing approach that recently introduced as alternative for interscalene brachial plexus nerve block in shoulder surgery. However, some researchers reported that Suprascapular nerve block alone results in an ineffective analgesia. Erector Spinae Plane block is supposed to be able in providing adequate analgesia in shoulder surgery

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II,
* Age above 21 years and below 60 years in both sexes,
* Cooperative patients,
* Patients with a BMI (body mass index) not exceeding 35.

Exclusion Criteria:

* patients with cardiovascular or respiratory compromise,
* Patient refusal,
* Coagulopathy,
* Local tissue infection,
* Allergy to local anesthesia,
* prior to cervical or thoracic spine surgery.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Intraoperative analgesia | The intraoperative patients' hemodynamics every 30 min were collected and analyzed till the end of surgery . Also the total dose of opioids consumed intraoperatively will be recorded. Postoperative consumed opioid for 24 hours also will calculated
  Recording of the patients' hemodynamics (heart rate and non-invasive blood pressure) and total dose of opioids consumption intraoperatively and postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available when the study is finished and the paper is published
Supporting Information: Study Protocol, SAP, CSR
Time Frame: once the paper is published and become available online
Access Criteria: for all anaesthesiologists
URL: https://www.clinicaltrials.gov/ct2/home

REFERENCES:
- [Background] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Background] Ma W, Sun L, Ngai L, Costouros JG, Steffner R, Boublik J, Tsui BCH. Motor-sparing high-thoracic erector spinae plane block for proximal humerus surgery and total shoulder arthroplasty surgery: clinical evidence for differential peripheral nerve block? Can J Anaesth. 2019 Oct;66(10):1274-1275. doi: 10.1007/s12630-019-01442-4. Epub 2019 Jul 9. No abstract available. PMID 31290120
- [Background] Hussain N, Goldar G, Ragina N, Banfield L, Laffey JG, Abdallah FW. Suprascapular and Interscalene Nerve Block for Shoulder Surgery: A Systematic Review and Meta-analysis. Anesthesiology. 2017 Dec;127(6):998-1013. doi: 10.1097/ALN.0000000000001894. PMID 28968280
- [Derived] Abdelhaleem NF, Abdelatiff SE, Abdel Naby SM. Comparison of Erector Spinae Plane Block at the Level of the Second Thoracic Vertebra With Suprascapular Nerve Block for Postoperative Analgesia in Arthroscopic Shoulder Surgery. Pain Physician. 2022 Nov;25(8):577-585. PMID 36375187